CLINICAL TRIAL: NCT05904301
Title: Armenian Nationwide Registry of Systemic Autoimmune and Autoinflammatory Diseases
Acronym: NAREG
Status: Recruiting | Type: Observational
Sponsor: Santé Arménie French-Armenian Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: SA-2021001
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2024-11

CONDITIONS: Behcet Disease; Antineutrophil Cytoplasmic Antibody (ANCA) Positive Vasculitis; Takayasu Arteritis; Giant Cell Arteritis; Sjogren's Syndrome; Rheumatoid Arthritis; Hereditary and Acquired Angioedema; Primary Antiphospholipid Syndrome; Celiac Disease
Keywords: arthritis; autoimmune; systemic; autoinflammatory; Behcet; Takayasu; Giant Cell; Angioedema; APS
MeSH Terms: conditions — Behcet Syndrome; Takayasu Arteritis; Giant Cell Arteritis; Sjogren's Syndrome; Arthritis, Rheumatoid; Acquired angioedema; Celiac Disease; Arthritis; Angioedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples (or components of the samples, PBMCs, DNA, serum, microbiota) taken as part of the study will be stored in a biological sample collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Systemic autoimmune and autoinflammatory diseases
  Interventions: Other: Usual medical management of patients, additional blood and stool samples for biobanking

INTERVENTIONS:
Other: Usual medical management of patients, additional blood and stool samples for biobanking — For all systemic diseases the following data will be collected:
  Clinical examination, Laboratory data, Current medications, Constitution of biobanking.
  For each disease:
  Pathology specific Activity score, Global subjective disease activity by patient and by physician.

SUMMARY:
Longitudinal prospective multicenter Armenian registry of systemic autoimmune, autoinflammatory diseases with constitution of bio-banking.

DETAILED DESCRIPTION:
Autoimmune and auto inflammatory diseases are a growing group of disorders caused by a dysregulation of the innate immune system leading to episodes of systemic inflammation.

They represent a group of diseases characterized by excessive autoimmune or inflammatory reaction leading to various organ damage and drop in patient's quality of life, usually underlined by particular genetic factors and environmental triggers.

The progress of these diseases is often evaluated in the form of activity scores.

A number of scores are available to predict the evolution of autoimmune autoinflammatory diseases.

For a long time, these pathologies have remained slightly explored because of their complex physiopathology and the absence of specific therapies.

In the last few years, significant progress has been made in terms of both pathophysiology and treatment.

Treatment with biological targeted therapies transformed the prognosis and survival of the patients, improved their quality of life and underlined the necessity of a global management of these patients.

In Armenia, the epidemiological elements of these pathologies are not known, nor are the circumstances of their discovery. The initial biological manifestations and the management of these patients are variable from one center to another, whether in terms of supportive or specific therapeutic elements.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of at least one of following autoimmune systemic diseases:

   Behcet disease, ANCA -positive vasculitis, Takayasu arteritis, Giant cell arteritis, Systemic sclerosis, Sjogren syndrome, Rheumatoid arthritis, Spondylarthritis (psoriatic, ankylosing, crohn's related), Angioedema hereditary and acquired, Pediatric dermatology, Autoinflammatory diseases (hereditary and acquired), Unexplained infertility, Immune thrombocytopenic purpura/ Autoimmune hemolytic anemia (ITP, AHA), Primary anti-phospholipid syndrome (APS), Celiac disease.
2. Age: major and minor
3. Patients who have been informed and provided with written informed consent to participate Or consent from legal representative

Exclusion Criteria:

1. Patients refusing to participate in the registry
2. Non-consent from legal representative
3. Breastfeeding or pregnant patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients and inpatients at participating centers, major and minor patients with a confirmed diagnosis of at least one of autoimmune systemic diseases
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Systemic manifestations and evolution of the diseases under treatment by disease-specific activity scores | Through study completion, an average of 5 years
  Description of Initial manifestations and the progress of these diseases.
  The progress of these diseases is assessed in the form of disease-specific activity scores:
  * ANCA-positive vasculitis - BVAS
  * Takayasu arthritis - NIH criteria
  * Rheumatoid arthritis - DAS28
  * Sjogren syndrome - ESSDAI, ESSRPI

SECONDARY OUTCOMES:
Identification of rare clinical forms | Through study completion, an average of 5 years
  Clinical and biological correlations to characterize rare clinical forms of each pathology
Prognostic factors of the diseases | Through study completion, an average of 5 years
  Interest in prognostic factors obtained through more targeted radiological examinations and correlation with the response to different treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Merry Mazmanian, Dr., Study Director — Santé Arménie French - Armenian Academic Research Organization FAARO
Locations (6):
- Armenia (6):
  - Hematology Center after Prof.R.H. Yeolyan, Yerevan
  - Nairi Medical Center, Rheumatology Department, Yerevan
  - Heratsi Hospital Complex n°1, Rheumatology Department, Yerevan
  - Heratsi Hospital Complex №1, Allergology Department, Yerevan
  - Mikaelyan Institute of Surgery, Rheumatology Department, Yerevan
  - Erebouni Medical Center, Rheumatology Department, Yerevan

IPD SHARING:
Plan to Share IPD: Undecided